CLINICAL TRIAL: NCT00463346
Title: Treatment With Acamprosate in Patients With Schizophrenia and Comorbid Alcoholism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0607001674; 0607001674; IP00027
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2015-12

CONDITIONS: Alcohol Dependence; Schizophrenia
Keywords: Treatment; Alcohol Dependence; Schizophrenia
MeSH Terms: conditions — Alcoholism; Schizophrenia | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acamprosate (Experimental): Acamprosate
  Interventions: Drug: Acamprosate
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acamprosate — Acamprosate 1998 mg tid
  Other Names: Campral
  Arms: Acamprosate
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of acamprosate for patients with alcohol dependence and comorbid schizophrenia spectrum disorders.

* 1: Relative to placebo, acamprosate will significantly increase cumulative days of abstinence in recently detoxified alcohol dependent schizophrenia patients measured by Timeline Follow-Back (TLFB) method.
* 2: Acamprosate will have no significant effect on the psychotic symptoms in schizophrenia patients with alcohol dependence as measured by the Positive and Negative Syndrome Scale (PANSS).

DETAILED DESCRIPTION:
Alcohol use disorders (AUD) are common comorbid conditions in patients with schizophrenia, and they cause a negative impact on the expression and course of schizophrenia. Improvements have been reported after attaining abstinence from alcohol, suggesting that effective treatments for AUD lead to clinically meaningful results. Acamprosate is a recently approved treatment for alcoholism, and it may be advantageous over other treatments since is not metabolized in the liver, and it has been used safely with other psychotropic medications. Therefore, acamprosate would be a promising treatment in schizophrenia patients. However, there are only few reports in the current literature evaluating the efficacy of medications available for the treatment of alcoholism in patients with schizophrenia, and the efficacy and safety of acamprosate have never been studied in this vulnerable group of patients.

Research Design:

This is a 12-week, randomized, double blind, placebo controlled trial of acamprosate (666 mg tid) in addition to neuroleptics in 30 recently abstinent (>5 days) schizophrenia patients with comorbid alcohol dependence.

Methods:

The study will be conducted at the West Haven, CT VA with support from Forest Laboratories. Patients who are between 21 and 65, with a diagnosis of schizophrenia spectrum disorder, (on stable psychotropic treatment > 2 weeks) and with current alcohol dependence (>1 recent episode of heavy drinking) will be included. Patients will be willing to undergo detoxification or self discontinuation >2weeks prior to the randomization. Main outcome variables include the TLFB method to document the degree of daily alcohol consumption, and PANSS, to assess the psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria

1. Men and women between 21 and 65 years of age.
2. Patients with a diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder NOS as determined by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID) [22].
3. Patients who are on stable treatment with psychotropic medication > 2 weeks prior to randomization.
4. Patients with current alcohol dependence, with at least one recent episode of heavy drinking (defined as 5 or more drinks per drinking episode) over the past 21 days, and willing to undergo detoxification or self discontinuation (for at least 5 days).
5. Patients, who are able to comprehend and satisfactorily comply with protocol requirements.
6. Patients who have capacity to provide informed consent prior to entering any study procedure.

Exclusion Criteria

1. Patients with dementia, amnestic and other cognitive disorders.
2. Patients who have unstable medical disease or a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial
3. Patients with a history of opioid dependence within the past month.
4. Patients with a history of intolerance or hypersensitivity to acamprosate.
5. Patients who are currently taking disulfiram or naltrexone.
6. Patients who based on history or mental status examination are at a significant risk for suicide.
7. Patients who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
8. Women who are pregnant or nursing, or women of childbearing potential who are sexually active and who do not use adequate contraception, or who are judged to be unreliable in their use of contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acamprosate: Acamprosate 1998 mg TID dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
- Placebo: dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 12 | 11
Completed | 9 | 8
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Individuals with schizophrenia, schizoaffective or psychotic disorder not otherwise specified and current alcohol dependence
Groups:
- Placebo: Placebo dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.27 (9.24) | 49.18 (4.64) | 50.73 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Acamprosate: Acamprosate
  1998 mg TID Study medication was dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
- Placebo: Placebo Study medication was dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 12 | 11
days | 10.7 (17.11) | 7.6 (11.5)

2. Primary Outcome: Psychotic Symptoms - Measured Using the PANSS
Description: The PANSS or the Positive and Negative Syndrome Scale is a medical scale used for measuring symptom severity of patients with schizophrenia. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale.The scores for these scales are arrived at by summation of ratings across component items. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. A higher score indicates more severe symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Acamprosate: Acamprosate
  Acamprosate: Acamprosate 1998 mg tid. Study medication was dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 12 | 11
units on a scale
  PANSS positive symptoms | 14.514 (1.263) | 14.362 (1.352)
  PANSS negative symptoms | 13.476 (1.388) | 15.971 (1.790)
  PANSS general symptoms | 28.083 (2.179) | 29.33 (2.345)

ADVERSE EVENTS:
Groups:
- Acamprosate: Acamprosate 1998 mg tid. Study medication was dispensed weekly in blister packs, labeled with the date and time, in identical looking capsules.
Arm/Group | Acamprosate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=12) | Placebo (N=11)
Hospitalized for fainting and vomiting (General disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization for psychiatric symptoms (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No